CLINICAL TRIAL: NCT04687072
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and the Safety of Efgartigimod (ARGX-113) PH20 Subcutaneous in Adult Patients With Primary Immune Thrombocytopenia
Brief Title: A Study to Evaluate the Efficacy and Safety of Efgartigimod PH20 Subcutaneous in Adult Patients With Primary Immune Thrombocytopenia
Acronym: ADVANCE SC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2004; 2020-004032-21 (EudraCT Number)
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod PH20 SC (Experimental): Patients receiving efgartigimod PH20 SC treatment
  Interventions: Biological: Efgartigimod PH20 SC
- Placebo PH20 SC (Placebo Comparator): Patients receiving placebo PH20 SC treatment
  Interventions: Other: Placebo PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous injection with efgartigimod PH20 SC
  Other Names: ARGX-113 PH20 SC
  Arms: Efgartigimod PH20 SC
Other: Placebo PH20 SC — Subcutaneous injection with placebo PH20 SC
  Arms: Placebo PH20 SC

SUMMARY:
This is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group trial to evaluate the efficacy, safety, and effect on QoL/PRO of efgartigimod PH20 SC treatment in adult patients with primary ITP.

ELIGIBILITY:
Inclusion criteria:

* Ability to understand the requirements of the trial and provide written informed consent, willing and able to comply with the trial protocol procedures
* Is at least the local age of consent for clinical studies when signing the ICF.
* Confirmed diagnosis of primary ITP made at least 3 months before randomization and based on the American Society of Hematology Criteria, and no known etiology for thrombocytopenia
* Diagnosis supported by a response to a prior ITP therapy (other than TPO-RAs), in the opinion of the investigator
* Mean platelet count of <30×10E9/L from at least 3 documented, qualifying counts within the 3 preceding months where at least 2 of the qualifying counts must be taken during the screening period: 1 platelet count collected during the screening period and the predose platelet count on the day of randomization (visit 1). If the third count is not available from the 3 preceding months, this third platelet count can be obtained during the screening period.
* A documented history of a platelet count of <30×10E9/L before screening
* At the start of the trial, the participant either takes concurrent ITP treatment(s) and has received at least 1 prior therapy for ITP in the past, or the participant does not take treatment for ITP (see note) but has received at least 2 prior treatments for ITP. Participants receiving permitted concurrent ITP treatment(s) at baseline must have been stable in dose and frequency for at least 4 weeks before randomization.

Permitted concurrent ITP medications include corticosteroids, danazol, vinca alkaloids, oral immunosuppressants, dapsone, fostamatinib, and/or oral TPO-RAs.

-Agree to use contraceptive measures consistent with local regulations and the protocol

Exclusion criteria:

* Secondary ITP/thrombocytopenia associated with another condition, eg, lymphoma, chronic lymphocytic leukemia, viral infection, hepatitis, induced or alloimmune thrombocytopenia, thrombocytopenia associated with myeloid dysplasia, or hematopoietic stem cell transplant
* Use of anticoagulants (eg, vitamin K antagonists, direct oral anticoagulants) within 4 weeks prior to randomization
* Use of any transfusions within 4 weeks prior to randomization
* Use of Ig (IV, SC, or intramuscular route) or plasmapheresis (PLEX) within 4 weeks prior to randomization
* Use of romiplostim within 4 weeks prior to randomization
* Undergone splenectomy less than 4 weeks prior to randomization
* Use of an investigational product within 3 months or 5 half-lives (whichever is longer) before the first dose of the IMP
* Use of any monoclonal antibody or Fc fusion proteins, other than those previously indicated, within 6 months before the first dose of the IMP (eg, anti-CD20)
* At the screening visit, clinically significant laboratory abnormalities as follows: Hemoglobin ≤9 g/dL - OR - International normalized ratio >1.5 or activated partial thromboplastin time >1.5×upper limit of normal - OR - total IgG level <6 g/L
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of IMP. Participants with the following cancer can be included at any time: Adequately treated basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast or Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
* Uncontrolled hypertension, defined as a repeated elevated blood pressure exceeding 160 mmHg (systolic) and/or 100 mmHg (diastolic) despite appropriate treatments
* History of any major thrombotic or embolic event (eg, myocardial infarction, stroke, deep venous thrombosis, or pulmonary embolism) within 5 years prior to randomization
* History of coagulopathy or hereditary thrombocytopenia or a family history of thrombocytopenia
* Evidence of an active clinically significant bleeding of an organ or internal mucosal bleeding, other than expected in ITP, that warrants emergent treatment or therapeutic procedure based on the investigator's judgment (eg, intracranial hemorrhage, pulmonary hemorrhage, bleeding with ongoing need for packed red blood cell transfusion)
* Estimated high risk of a clinically significant bleeding of an organ or internal mucosal bleeding, other than expected in ITP, that warrants emergent treatment or therapeutic procedure according to the investigator's judgment
* Clinical evidence of other significant serious diseases, have had a recent major surgery, or who have any other condition in the opinion of the investigator, that could confound the results of the trial or put the participant at undue risk
* Positive serum test at screening for an active viral infection with any of the following conditions: Hepatitis B virus (HBV) that is indicative of an acute or chronic infection, unless associated with a negative HBV DNA test, Hepatitis C virus (HCV) based on HCV-antibody assay (unless associated with a negative HCV RNA test), Human immunodeficiency virus (HIV) based on test results that are associated with an acquired immunodeficiency syndrome (AIDS)-defining condition or a CD4 count ≤200 cells/mm3
* Known hypersensitivity reaction to efgartigimod, rHuPH20, or 1 of its excipients
* Previously participated in a clinical trial with efgartigimod and have received at least 1 administration of the IMP
* Pregnant or lactating or intends to become pregnant during the trial
* Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening
* Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of ITP or put the participant at undue risk
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases other than ITP (eg, cardiovascular, pulmonary, hematologic, gastrointestinal, endocrine, hepatic, renal, neurological, malignancy, infectious diseases, uncontrolled diabetes) despite appropriate treatments which could put the participant at undue risk
* Current or history of (ie, within 12 months of screening) alcohol, drug, or medication abuse
* Received a live/live-attenuated vaccine less than 4 weeks before screening. The receipt of any inactivated, sub-unit, polysaccharide, or conjugate vaccine at any time before screening is not considered an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (200):
- United States (14):
  - Investigator Site 0010116, Springdale, Arkansas
  - Investigator site 0010036, Los Angeles, California
  - Investigator Site 0010045, Washington D.C., District of Columbia
  - Investigator Site 0010104, Weston, Florida
  - Investigator site 0010112, Chicago, Illinois
  - Investigator site 0010193, Chicago, Illinois
  - Investigator Site 0010079, Lisle, Illinois
  - Investigator Site 0010062, Fort Wayne, Indiana
  - Investigator site 0010042, Iowa City, Iowa
  - Investigator Site 0010083, Detroit, Michigan
  - Investigator Site 0010102, Minneapolis, Minnesota
  - Investigator site 0010040, Columbus, Ohio
  - Investigator Site 0010095, Oklahoma City, Oklahoma
  - Investigator Site 0010115, Pittsburgh, Pennsylvania
- Argentina (3):
  - Investigator Site 0540001, Buenos Aires
  - Investigator Site 0540004, Buenos Aires
  - Investigator Site 0540003, Córdoba
- Australia (9):
  - Investigator Site 0610009, Adelaide
  - Investigator Site 0610004, Bedford Park
  - Investigator Site 0610002, Box Hill
  - Investigator Site 0610010, Clayton
  - Investigator Site 0610012, Garran
  - Investigator Site 0610001, Hobart
  - Investigator Site 0610011, Perth
  - Investigator Site 0610003, West Perth
  - Investigator Site 0610005, Westmead
- Bulgaria (2):
  - Investigator Site 3590017, Plovdiv
  - Investigator Site 3590015, Sofia
- Chile (3):
  - Investigator Site 0560002, Santiago
  - Investigator Site 0560004, Temuco
  - Investigator Site 0560003, Viña del Mar
- China (16):
  - Investigator Site 0860003, Beijing
  - Investigator Site 0860013, Beijing
  - Investigator Site 0860008, Bengbu
  - Investigator Site 0860055, Huizhou
  - Investigator Site 0860009, Kunming
  - Investigator Site 0860012, Nanchang
  - Investigator Site 0860014, Shanxi
  - Investigator Site 0860015, Shenzhen
  - Investigator Site 0860001, Tianjin
  - Investigator Site 0860006, Wenzhou
  - Investigator Site 0860010, Wuhan
  - Investigator Site 0860002, Wuxi
  - Investigator Site 0860005, Zhejiang
  - Investigator Site 0860011, Zhengzhou
  - Investigator Site 0860058, Zhenjiang
  - Investigator site 0860062, Zhenjiang
- Investigator Site 0450005, Roskilde, Denmark
- France (2):
  - Investigator Site 0330009, Créteil
  - Investigator Site 0330018, Montpellier
- Georgia (6):
  - Investigator Site 9950006, Tbilisi
  - Investigator Site 9950007, Tbilisi
  - Investigator Site 9950008, Tbilisi
  - Investigator Site 9950009, Tbilisi
  - Investigator Site 9950011, Tbilisi
  - Investigator Site 9950019, Tbilisi
- Germany (2):
  - Investigator site 0490008, Essen
  - Investigator Site 0490012, Giessen
- Greece (4):
  - Investigator Site 0300008, Athens
  - Investigator Site 0300010, Athens
  - Investigator Site 0300007, Pátrai
  - Investigator Site 0300009, Thessaloniki
- Ireland (3):
  - Investigator Site 3530002, Dublin
  - Investigator Site 3530003, Dublin
  - Investigator Site 3530001, Galway
- Israel (7):
  - Investigator Site 9720013, Ashkelon
  - Investigator Site 9720010, Haifa
  - Investigator Site 9720012, Haifa
  - Investigator Site 9720008, Jerusalem
  - Investigator Site 9720011, Jerusalem
  - Investigator Site 9720007, Petah Tikva
  - Investigator Site 9720009, Tel Aviv
- Italy (14):
  - Investigator Site 0390037, Alessandria
  - Investigator Site 0390043, Ferrara
  - Investigator Site 0390045, Meldola
  - Investigator site 0390014, Milan
  - Investigator Site 0390032, Milan
  - Investigator Site 0390041, Napoli
  - Investigator Site 0390044, Napoli
  - Investigator Site 0390015, Novara
  - Investigator Site 0390035, Potenza
  - Investigator Site 0390011, Reggio Calabria
  - Investigator site 0390018, Reggio Emilia
  - Investigator Site 0390046, Rome
  - Investigator Site 0390033, Terni
  - Investigator Site 0390036, Varese
- Japan (17):
  - Investigator Site 0810056, Chiba
  - Investigator Site 0810015, Hirakata
  - Investigator Site 0810010, Hiroshima
  - Investigator Site 0810053, Kanagawa
  - Investigator Site 0810051, Kitakyushu
  - Investigator Site 0810054, Kumamoto
  - Investigator Site 0810018, Maebashi
  - Investigator Site 0810057, Morioka
  - Investigator Site 0810012, Ōgaki
  - Investigator Site 0810017, Saitama
  - Investigator Site 0810016, Shibukawa
  - Investigator Site 0810023, Shimotsuke
  - Investigator Site 0810039, Shinagawa-Ku
  - Investigator Site 0810038, Tama
  - Investigator Site 0810052, Tokyo
  - Investigator Site 0810048, Tsukuba
  - Investigator Site 0810044, Yamanashi
- Jordan (2):
  - Investigator Site 9620002, Amman
  - Investigator Site 9620001, Irbid
- Mexico (5):
  - Investigator Site 0520002, Aguascalientes
  - Investigator Site 0520004, Chihuahua City
  - Investigator Site 0520007, México
  - Investigator Site 0520003, Monterrey
  - Investigator Site 0520001, Oaxaca City
- New Zealand (3):
  - Investigator Site 0640001, Auckland
  - Investigator Site 0640005, Christchurch
  - Investigator Site 0640002, Palmerston North
- Norway (2):
  - Investigator Site 0470002, Bergen
  - Investigator Site 0470003, Oslo
- Poland (6):
  - Investigator Site 0480013, Katowice
  - Investigator Site 0480014, Lublin
  - Investigator Site 0480026, Nowy Sącz
  - Investigator Site 0480037, Skorzewo
  - Investigator Site 0480039, Torun
  - Investigator Site 0480033, Warsaw
- Portugal (7):
  - Investigator Site 3510006, Braga
  - Investigator Site 3510003, Coimbra
  - Investigator Site 3510002, Lisbon
  - Investigator Site 3510005, Lisbon
  - Investigator Site 3510007, Lisbon
  - Investigator Site 3510001, Porto
  - Investigator Site 3510004, Porto
- Romania (8):
  - Investigator Site 0400005, Bucharest
  - Investigator Site 0400006, Bucharest
  - Investigator Site 0400009, Bucharest
  - Investigator Site 0400012, Bucharest
  - Investigator Site 0400016, Cluj-Napoca
  - Investigator Site 0400007, Craiova
  - Investigator Site 0400011, Sibiu
  - Investigator Site 0400008, Târgu Mureş
- Russia (10):
  - Investigator Site 0070006, Kaluga
  - Investigator Site 0070040, Kirov
  - Investigator Site 0070026, Moscow
  - Investigator Site 0070038, Nizhny Novgorod
  - Investigator Site 0070037, Novosibirsk
  - Investigator Site 0070024, Pyatigorsk
  - Investigator Site 0070025, Saint Petersburg
  - Investigator Site 0070039, Smolensk
  - Investigator Site 0070015, Syktyvkar
  - Investigator Site 0070012, Tula
- Serbia (2):
  - Investigator Site 3810006, Belgrade
  - Investigator Site 3810008, Kragujevac
- South Africa (5):
  - Investigator Site 0270005, George
  - Investigator Site 0270003, Johannesburg
  - Investigator Site 0270004, Observatory
  - Investigator Site 0270001, Pretoria
  - Investigator Site 0270002, Randburg
- South Korea (6):
  - Investigator Site 0820005, Seongnam
  - Investigator Site 0820003, Seoul
  - Investigator Site 0820004, Seoul
  - Investigator Site 0820006, Seoul
  - Investigator Site 0820007, Seoul
  - Investigator Site 0820008, Seoul
- Spain (9):
  - Investigator Site 0340024, Alava
  - Investigator Site 0340007, Barcelona
  - Investigator Site 0340006, Barcelona
  - Investigator Site 0340023, Barcelona
  - Investigator Site 0340037, Madrid
  - Investigator Site 0340022, Murcia
  - Investigator Site 0340036, Sabadell
  - Investigator site 0340013, Seville
  - Investigator Site 0340004, Valencia
- Taiwan (2):
  - Investigator Site 8860001, New Taipei City
  - Investigator Site 8860003, Taoyuan District
- Thailand (8):
  - Investigator Site 0660002, Bangkok
  - Investigator Site 0660003, Bangkok
  - Investigator Site 0660005, Bangkok
  - Investigator Site 0660008, Bangkok
  - Investigator Site 0660001, Bangkok Noi
  - Investigator Site 0660004, Chiang Mai
  - Investigator Site 0660009, Khon Kaen
  - Investigator Site 0660006, Pathum Thani
- Tunisia (3):
  - Investigator Site 2160006, Sfax
  - Investigator Site 2160001, Sousse
  - Investigator Site 2160002, Tunis
- Turkey (Türkiye) (14):
  - Investigator Site 0900007, Adapazarı
  - Investigator Site 0900003, Ankara
  - Investigator Site 0900006, Ankara
  - Investigator Site 0900008, Ankara
  - Investigator Site 0900015, Ankara
  - Investigator Site 0900016, Edirne
  - Investigator Site 0900013, Istanbul
  - Investigator Site 0900004, Izmir
  - Investigator Site 0900014, Kocaeli
  - Investigator Site 0900018, Malatya
  - Investigator Site 0900010, Mersin
  - Investigator Site 0900009, Samsun
  - Investigator Site 0900017, Tekirdağ
  - Investigator Site 0900019, Trabzon
- United Kingdom (5):
  - Investigator site 0440011, Bradford
  - Investigator Site 0440005, Coventry
  - Investigator Site 0440008, London
  - Investigator Site 0440041, London
  - Investigator Site 0440014, Truro

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A regionally diverse participant population was enrolled (including but not limited to North America, East Asia, Europe, and the rest of world [ROW]).
  A total of 207 participants were randomized to IMP: 137 participants in the efgartigimod PH20 subcutaneous (SC) arm and 70 participants in the placebo PH20 SC arm.
Groups:
- Efgartigimod PH20 SC: Participants receiving efgartigimod PH20 SC treatment.
- Placebo PH20 SC: Participants receiving placebo PH20 SC treatment.
Period: Overall Study
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Started | 137 | 70
Completed | 113 | 62
Not Completed | 24 | 8
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Requires Prohibited Medication | 2 | 0
Not completed — Withdrawal of Consent | 11 | 6
Not completed — Miscellaneous | 4 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): All participants who received at least 1 dose or part of a dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC | Total
Number analyzed (Participants) | 137 | 70 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (17.22) | 50.0 (15.29) | 48.2 (16.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 43 | 131
  Male | 49 | 27 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 129 | 68 | 197
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 44 | 18 | 62
  Black or African American | 4 | 2 | 6
  White | 88 | 49 | 137
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Chronic Immune Thrombocytopenia (ITP) With a Sustained Platelet Count Response Between Weeks 19 and 24
Description: A participant was considered a responder for this endpoint (i.e., had a sustained platelet count response) if the participant had platelet counts of ≥50 × 10^9/L for ≥4 of the 6 analysis visits between Weeks 19 and 24.
Time Frame: Up to 6 weeks (between Weeks 19 and 24)
Population: Full Analysis Set (FAS)-Chronic: Participants from the FAS (all randomized participants) including only participants with chronic ITP.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 68
percentage of participants | 13.7 | 16.2
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.5081, Cochran-Mantel-Haenszel — The p-value was calculated using the Cochran-Mantel-Haenszel test used in the hierarchical testing procedure; Difference in percentage = -3.5, 95% CI 2-sided [-14.7 to 7.0] — The adjusted difference in percentages and 95% confidence interval (CI) (Klingenberg approach) were presented

2. Secondary Outcome: Extent of Disease Control Over the 24-Week Treatment Period in the Chronic ITP Population
Description: Extent of disease control was defined as the number of cumulative weeks over the planned 24-week treatment period with platelet counts of ≥50×10^9/L in the chronic ITP population.
Time Frame: Up to 24 weeks
Population: FAS-Chronic: Participants from the FAS (all randomized participants) including only participants with chronic ITP.
Measure: Median (Full Range); unit: weeks
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 68
weeks | 0.5 [0 to 24] | 0.0 [0 to 23]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.4925, Wilcoxon (Mann-Whitney) — The p-value was calculated using the stratified Mann-Whitney test used in the hierarchical testing procedure; Location shift = 0.000, 95% CI 2-sided [0.000 to 0.000] — The Hodges-Lehmann estimator of the treatment difference and 95% CI are presented

3. Secondary Outcome: Percentage of Participants in the Overall Population (Chronic and Persistent ITP) With a Sustained Platelet Count Response Between Weeks 19 and 24
Description: as for outcome 1
Time Frame: Up to 6 weeks (between Weeks 19 and 24)
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants | 16.1 | 15.7
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.9314, Cochran-Mantel-Haenszel — The p-value was calculated using the Cochran-Mantel-Haenszel test used in the hierarchical testing procedure; Difference in percentage = -0.5, 95% CI 2-sided [-11.7 to 10.0] — The adjusted difference in percentages and 95% CI (Klingenberg approach) were presented

4. Secondary Outcome: Percentage of Participants in the Overall Population With Sustained Platelet Count Response Between Weeks 17 and 24
Description: A participant was considered a responder for this endpoint (i.e., had a sustained platelet count response) if the participant had platelet counts of ≥50 × 10^9/L for ≥6 of the 8 analysis visits between weeks 17 and 24.
Time Frame: Up to 8 weeks (between Weeks 17 and 24)
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants | 12.4 | 14.3
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.7379, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel test p-value was used in the hierarchical testing procedure; Difference in percentage = -1.7, 95% CI 2-sided [-12.4 to 8.2] — The adjusted difference in percentage and 95% CI (Klingenberg approach) are presented

5. Secondary Outcome: Percentage of Participants in the Overall Population Achieving Overall Platelet Count Response at Any Time During the 24-week Treatment Period
Description: A participant was considered a responder for this endpoint (i.e., had an overall platelet count response) if the participant had platelet counts of ≥50 × 10^9/L for ≥4 analysis visits at any time during the 24-week treatment period.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants | 29.9 | 25.7
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Other; Difference in percentage = 4.2, 95% CI 2-sided [-9.3 to 16.8]; The 95% Agresti-Min CIs are presented

6. Secondary Outcome: Extent of Disease Control Until Week 12 in the Overall Population
Description: Extent of disease control was defined as the number of cumulative weeks until Week 12 with platelet counts of ≥50×10^9/L in the overall population.
Time Frame: Up to 12 weeks
Population: FAS: All randomized participants.
Measure: Median (Full Range); unit: weeks
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
weeks | 0.00 [0.00 to 12.00] | 0.00 [0.00 to 11.00]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.7260, Wilcoxon (Mann-Whitney) — The p-value was calculated using the stratified Mann-Whitney test; Location shift = 0.000, 95% CI 2-sided [0.000 to 0.000] — The Hodges-Lehmann estimator of the treatment difference and 95% CI are presented

7. Secondary Outcome: Percentage of Participants in the Overall Population Achieving Overall Platelet Count Response at Any Time Until Week 12
Description: A participant was considered a responder for this endpoint (i.e., had an overall platelet count response) if the participant had platelet counts of ≥50 × 10^9/L for ≥4 analysis visits at any time until Week 12.
Time Frame: Up to 12 weeks
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants | 18.2 | 15.7
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Other; Difference in percentage = 2.5, 95% CI 2-sided [-9.6 to 13.0] — The 95% Agresti-Min CIs are presented

8. Secondary Outcome: Mean Change From Baseline in Platelet Count at Each Visit in the Overall Population
Description: Change from Baseline at time point t = value at time point t - Baseline value. Baseline was defined as the last available value prior to first administration of the investigational medicinal product (IMP).
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, Safety and Efficacy Follow-up Visit 1 (SEFU1) (up to Week 29), and SEFU2 (up to Week 33)
Population: FAS: All randomized participants with available data.
Measure: Mean (Standard Deviation); unit: platelets x10^9/L
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 136 | 69
platelets x10^9/L
  Week 1 | 13.84 (41.150) | 8.82 (34.355)
  Week 2: number analyzed (Participants) | 135 | 68
  Week 2 | 16.62 (49.408) | 23.54 (85.005)
  Week 3: number analyzed (Participants) | 133 | 69
  Week 3 | 17.07 (39.855) | 19.22 (71.947)
  Week 4: number analyzed (Participants) | 132 | 68
  Week 4 | 12.39 (37.886) | 9.31 (26.813)
  Week 5: number analyzed (Participants) | 129 | 67
  Week 5 | 18.14 (54.335) | 12.24 (30.059)
  Week 6: number analyzed (Participants) | 127 | 65
  Week 6 | 34.61 (112.204) | 16.35 (40.891)
  Week 7: number analyzed (Participants) | 126 | 67
  Week 7 | 28.25 (107.932) | 13.46 (41.876)
  Week 8: number analyzed (Participants) | 126 | 66
  Week 8 | 21.77 (52.308) | 16.57 (42.508)
  Week 9: number analyzed (Participants) | 123 | 64
  Week 9 | 19.90 (54.542) | 20.42 (53.488)
  Week 10: number analyzed (Participants) | 119 | 66
  Week 10 | 21.73 (47.685) | 15.42 (33.119)
  Week 11: number analyzed (Participants) | 122 | 63
  Week 11 | 20.13 (42.193) | 14.54 (25.588)
  Week 12: number analyzed (Participants) | 120 | 62
  Week 12 | 21.02 (43.882) | 22.28 (56.173)
  Week 13: number analyzed (Participants) | 118 | 63
  Week 13 | 22.29 (44.654) | 15.51 (37.651)
  Week 14: number analyzed (Participants) | 119 | 65
  Week 14 | 23.60 (47.521) | 24.04 (55.678)
  Week 15: number analyzed (Participants) | 116 | 59
  Week 15 | 21.30 (45.776) | 28.05 (67.897)
  Week 16: number analyzed (Participants) | 113 | 58
  Week 16 | 30.32 (71.553) | 23.09 (46.154)
  Week 17: number analyzed (Participants) | 112 | 58
  Week 17 | 25.12 (54.747) | 30.05 (56.581)
  Week 18: number analyzed (Participants) | 115 | 60
  Week 18 | 28.54 (53.115) | 31.64 (57.309)
  Week 19: number analyzed (Participants) | 114 | 62
  Week 19 | 33.86 (59.323) | 37.26 (68.832)
  Week 20: number analyzed (Participants) | 107 | 61
  Week 20 | 30.87 (55.342) | 25.85 (48.409)
  Week 21: number analyzed (Participants) | 108 | 59
  Week 21 | 30.04 (61.438) | 26.23 (50.323)
  Week 22: number analyzed (Participants) | 110 | 61
  Week 22 | 33.26 (61.558) | 29.23 (55.175)
  Week 23: number analyzed (Participants) | 111 | 60
  Week 23 | 29.51 (53.437) | 24.89 (41.103)
  Week 24: number analyzed (Participants) | 113 | 59
  Week 24 | 25.51 (52.203) | 24.91 (42.972)
  SEFU1: number analyzed (Participants) | 9 | 1
  SEFU1 | 40.44 (64.860) | 48.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  SEFU2: number analyzed (Participants) | 10 | 2
  SEFU2 | 30.00 (35.011) | 56.25 (85.206)

9. Secondary Outcome: Time to Platelet Count Response in the Overall Population
Description: Time to platelet count response, defined as the time to have 2 consecutive platelet counts of ≥50 × 10^9/L via Kaplan-Meier estimates.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants. Participants with no occurrence of platelet count response, early discontinuation of treatment, or dose and/or frequency of concurrent ITP therapy increased or a new ITP therapy were censored. If multiple censoring conditions apply, the earliest censoring date is considered.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
days | NA [155.0 to NA] — Median and upper confidence interval were not calculable due to fewer than 50% events. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient number of events.

10. Secondary Outcome: Extent of Disease Control Over the 24-Week Treatment Period in the Overall Population
Description: Extent of disease control was defined as the number of cumulative weeks over the planned 24-week treatment period with platelet counts of ≥30×10^9/L with at least ≥20×10^9/L above Baseline in the overall population.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants.
Measure: Median (Full Range); unit: weeks
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
weeks | 1.0 [0 to 24] | 1.0 [0 to 24]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.2929, Wilcoxon (Mann-Whitney) — The p-value was calculated using the stratified Mann-Whitney test; Location shift = 0.000, 95% CI 2-sided [0.000 to 1.000] — The Hodges-Lehmann estimator of the treatment difference and 95% CI are presented

11. Secondary Outcome: Extent of Disease Control Over the 24-Week Treatment Period in the Overall Population for Participants With Baseline Platelet Count of <15×10^9/L
Description: as for outcome 10
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants with Baseline Platelet Count of <15×10^9/L.
Measure: Median (Full Range); unit: weeks
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 59 | 35
weeks | 1.0 [0 to 23] | 0.0 [0.0 to 24]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Superiority; p = 0.1475, Wilcoxon (Mann-Whitney) — The p-value was calculated using the stratified Mann-Whitney test; Location shift = 0.000, 95% CI 2-sided [0.000 to 1.000] — The Hodges-Lehmann estimator of the treatment difference and 95% CI are presented

12. Secondary Outcome: Number of the World Health Organization (WHO)-Classified Bleeding Events (Grade ≥1) in the Overall Population
Description: Assessed using the WHO bleeding scale. The WHO bleeding scale is a five-point scale where Grade 0 = no bleeding; Grade 1 = petechial bleeding; Grade 2 = mild blood loss; Grade 3 = gross blood loss (requires transfusion); and Grade 4 = debilitating blood loss, associated with fatality.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants.
Measure: Median (Full Range); unit: bleeding events
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
bleeding events | 9.0 [0 to 24] | 10.0 [0 to 24]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; WHO Classified Bleeding Event Grade ≥1; Test type: Superiority; p = 0.7677, Wilcoxon (Mann-Whitney) — The p-value was calculated using the stratified Mann-Whitney test used in the hierarchical testing procedure; Location shift = 0.000, 95% CI 2-sided [-2.000 to 2.000] — The Hodges-Lehmann estimator of the treatment difference and 95% CI are presented

13. Secondary Outcome: Percentage of Participants With a Platelet Count International Working Group (IWG) Response
Description: IWG complete response was defined as platelet counts of ≥100 × 10^9/L and the absence of bleeding events (WHO Grading = 0 [no bleeding]) for at least 2 separate, consecutive analysis visits at least 7 days apart.
  IWG response was defined as platelet counts of ≥30 × 10^9/L and a 2-fold increase of platelet count from Baseline and the absence of bleeding events (WHO grading = 0) for at least 2 separate, consecutive analysis visits that were at least 7 days apart.
  Initial response was defined as platelet counts of ≥30 × 10^9/L and a 2-fold increase from the Baseline platelet count at analysis visit 5.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants
  IWG Complete Response | 10.2 | 11.4
  IWG Response | 28.5 | 20.0
  Initial Response | 19.7 | 17.1
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; IWG Complete Response; Test type: Other; Difference in percentage = -1.2, 95% CI 2-sided [-11.8 to 7.3] — The 95% Agresti-Min CIs are presented
Statistical Analysis 2: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; IWG Response; Test type: Other; Difference in percentage = 8.5, 95% CI 2-sided [-4.6 to 20.2] — The 95% Agresti-Min CIs are presented
Statistical Analysis 3: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Initial Response; Test type: Other; Difference in percentage = 2.6, 95% CI 2-sided [-9.7 to 13.3] — The 95% Agresti-Min CIs are presented

14. Secondary Outcome: Rate of Receipt of Rescue Therapy (Rescue Per Participant Per Month) in the Overall Population
Description: Rescue therapy was defined as an occurrence where the participant needed treatment with 1 or more rescue treatments. An occurrence was defined as a period of maximum 5 days where 1 or more rescue treatments were administered simultaneously or consecutively to the trial participant. The following rescue treatments were permitted: methylprednisolone, dexamethasone, prednisone, normal immunoglobulins, anti-D (Rho) immunoglobins, or platelet transfusions.
Time Frame: Up to 24 weeks
Population: FAS: All randomized participants.
Measure: Mean (Standard Deviation); unit: rescues per participant per month
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
rescues per participant per month | 0.25 (0.553) | 0.17 (0.363)

15. Secondary Outcome: Percentage of Participants for Whom Dose and/or Frequency of Concurrent ITP Therapies Have Increased at Week 12 or Later in the Overall Population
Description: A change in ITP therapy was defined as either an increase in the dose and/or frequency of a concurrent ITP therapy relative to Baseline or the initiation of a new concurrent ITP therapy.
Time Frame: Up to 13 weeks (between Weeks 12 and 24)
Population: FAS: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
percentage of participants | 11.7 | 15.7
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Placebo PH20 SC; Test type: Other; Difference in percentage = -4.0, 95% CI 2-sided [-15.6 to 5.7] — The 95% Agresti-Min CIs are presented

16. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-Fatigue) at Week 24 in the Overall Population
Description: The FACIT-fatigue scale is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during his/her usual daily activities over the past week. The level of fatigue was measured by recording item responses on a 5-point Likert scale ranging from 0 "not at all" to 4 "very much". All items were summed to create a single fatigue score with a range from 0 to 52, where a higher FACIT-F score indicated more severe symptoms. A negative change score from Baseline indicated improvement in quality of life (QoL).
Time Frame: Baseline and Week 24
Population: FAS: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
score on a scale | -0.025 (0.712) | 0.741 (0.985)

17. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy Questionnaire-Th6 (Fact-Th6) at Week 24 in the Overall Population
Description: The FACT-Th6 uses a 5-level Likert scale (0=not at all to 4=very much), with participants rating their degree of concern in the past 7 days. The 6 selected items pertain to ability to do usual activities, worry about problems with bleeding or bruising, worry about the possibility of serious bleeding, avoidance of physical or social activity because of concern with bleeding or bruising and frustration due to the inability to carry out usual activities. All items were summed to create a single score with a range from 0 to 24, where a higher score indicated less severe symptoms. A positive change score from Baseline indicated improvement in QoL.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: FAS: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
score on a scale | 0.225 (0.360) | 0.359 (0.498)

18. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) at Week 24 in the Overall Population
Description: The SF-36 is a 36-item scale constructed to survey health-related QoL on 8 domains: limitations in physical activities due to health problems; limitations in social activities due to physical or emotional problems; limitations in usual role activities due to physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities due to emotional problems; vitality (energy and fatigue); and general health perceptions. The scores from the 8 domains were evaluated independently and aggregated into 2 norm-based summary component measures of physical and mental health. The summary component scores could range from 0 to 100, where a higher score indicated improvement in QoL. A positive change score from Baseline indicated improvement in QoL.
Time Frame: Baseline and Week 24
Population: FAS: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 137 | 70
score on a scale
  Week 24: Mental Component | 1.215 (0.620) | 0.957 (0.841)
  Week 24: Physical Component | -0.848 (0.525) | -0.850 (0.712)

19. Secondary Outcome: Incidence and Prevalence of Antibodies to Efgartigimod and/or rHuPH20 in the Overall Population
Description: Anti-drug antibody (ADA) incidence was defined as the percentage of participants with treatment-induced or treatment boosted ADA (denominator: number of evaluable participants). ADA prevalence was defined as the percentage of participants with treatment-unaffected ADA, treatment-induced ADA or treatment-boosted ADA (denominator: number of evaluable participants).
Time Frame: Up to 35 weeks
Population: SAF: All participants who received at least 1 dose or part of a dose including only antibody-evaluable participants.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 136 | 70
percentage of participants
  Incidence of Antibodies to Efgartigimod | 5.1 | 2.9
  Prevalence of Antibodies to Efgartigimod | 16.2 | 7.1
  Incidence of Antibodies to rHuPH20 | 41.2 | 20.0
  Prevalence of Antibodies to rHuPH20 | 50.0 | 31.4

20. Secondary Outcome: Titers of Antibodies to Efgartigimod and/or rHuPH20 in the Overall Population
Description: A titer was determined in the samples with a positive assay response.
Time Frame: Weeks 3, 7, 11, 15, 19, 23, 24, SEFU1 (up to Week 29), and SEFU2 (up to Week 33)
Population: SAF: All participants who received at least 1 dose or part of a dose with available data.
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 45 | 16
titer
  Week 3: ADA Against Efgartigimod Titer: number analyzed (Participants) | 0 | 2
  Week 3: ADA Against Efgartigimod Titer |  | 16.5 (15.50)
  Week 7: ADA Against Efgartigimod Titer: number analyzed (Participants) | 1 | 3
  Week 7: ADA Against Efgartigimod Titer | 1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 11.3 (10.33)
  Week 11: ADA Against Efgartigimod Titer: number analyzed (Participants) | 0 | 3
  Week 11: ADA Against Efgartigimod Titer |  | 6.3 (4.84)
  Week 15: ADA Against Efgartigimod Titer: number analyzed (Participants) | 0 | 2
  Week 15: ADA Against Efgartigimod Titer |  | 8.5 (7.50)
  Week 19: ADA Against Efgartigimod Titer: number analyzed (Participants) | 0 | 0
  Week 23: ADA Against Efgartigimod Titer: number analyzed (Participants) | 0 | 1
  Week 23: ADA Against Efgartigimod Titer |  | 2.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Week 24: ADA Against Efgartigimod Titer: number analyzed (Participants) | 3 | 2
  Week 24: ADA Against Efgartigimod Titer | 16.3 (8.95) | 1.0 (0.00)
  SEFU1: ADA Against Efgartigimod Titer: number analyzed (Participants) | 2 | 0
  SEFU1: ADA Against Efgartigimod Titer | 2.5 (1.50) |
  SEFU2: ADA Against Efgartigimod Titer: number analyzed (Participants) | 2 | 0
  SEFU2: ADA Against Efgartigimod Titer | 17.0 (15.00) |
  Week 3: ADA Against rHuPH20 Titer: number analyzed (Participants) | 15 | 11
  Week 3: ADA Against rHuPH20 Titer | 12.7 (2.53) | 14.1 (3.15)
  Week 7: ADA Against rHuPH20 Titer: number analyzed (Participants) | 23 | 8
  Week 7: ADA Against rHuPH20 Titer | 645.9 (314.79) | 14.4 (4.27)
  Week 11: ADA Against rHuPH20 Titer: number analyzed (Participants) | 32 | 7
  Week 11: ADA Against rHuPH20 Titer | 2204.8 (1297.43) | 11.4 (2.37)
  Week 15: ADA Against rHuPH20 Titer: number analyzed (Participants) | 34 | 7
  Week 15: ADA Against rHuPH20 Titer | 3209.3 (1325.96) | 15.7 (2.02)
  Week 19: ADA Against rHuPH20 Titer: number analyzed (Participants) | 42 | 11
  Week 19: ADA Against rHuPH20 Titer | 3742.7 (1414.15) | 49.1 (27.87)
  Week 23: ADA Against rHuPH20 Titer: number analyzed (Participants) | 45 | 15
  Week 23: ADA Against rHuPH20 Titer | 5936.6 (2180.33) | 58.3 (27.83)
  Week 24: ADA Against rHuPH20 Titer | 4731.3 (1898.96) | 69.1 (26.60)
  SEFU1: ADA Against rHuPH20 Titer: number analyzed (Participants) | 2 | 0
  SEFU1: ADA Against rHuPH20 Titer | 5122.5 (5117.50) |
  SEFU2: ADA Against rHuPH20 Titer: number analyzed (Participants) | 2 | 0
  SEFU2: ADA Against rHuPH20 Titer | 5160.0 (5080.00) |

21. Secondary Outcome: Incidence and Prevalence of Neutralizing Antibodies (NAb) to Efgartigimod and/or rHuPH20 in the Overall Population
Description: Samples were tested for the presence of NAb against efgartigimod and/or rHuPH20 and titers for NAb against rHuPH20.
  NAb incidence is defined as the total percentage of participants with participant classification "baseline negative-postbaseline positive" and "baseline positive-postbaseline positive". NAb prevalence is defined as the total percentage of participants with participant classification "baseline negative-postbaseline positive," "baseline positive-postbaseline positive," or "baseline positive-postbaseline negative".
Time Frame: Up to 35 weeks
Population: SAF: All participants who received at least 1 dose or part of a dose with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 136 | 70
percentage of participants
  Incidence of NAb to Efgartigimod | 0.7 | 0.0
  Prevalence of NAb to Efgartigimod | 5.1 | 0.0
  Incidence of NAb to rHuPH20 | 0.0 | 0.0
  Prevalence of NAb to rHuPH20 | 0.0 | 0.0

22. Secondary Outcome: Serum Efgartigimod Trough Concentration (Ctrough) in the Overall Population
Description: All pharmacokinetic (PK) samples were collected predose, on the day of IMP administration.
Time Frame: Predose on Weeks 1, 2, 3, 17, 19, 21, 23, and 24
Population: PK Analysis Set: Safety analysis set excluding placebo participants and including participants with at least one serum post dose PK measurement.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 135
μg/mL
  Week 1 | 13.2 (6.46)
  Week 2: number analyzed (Participants) | 133
  Week 2 | 16.6 (8.17)
  Week 3: number analyzed (Participants) | 126
  Week 3 | 17.0 (7.95)
  Week 17: number analyzed (Participants) | 89
  Week 17 | 15.1 (8.54)
  Week 19: number analyzed (Participants) | 91
  Week 19 | 15.4 (7.43)
  Week 21: number analyzed (Participants) | 78
  Week 21 | 15.1 (8.86)
  Week 23: number analyzed (Participants) | 88
  Week 23 | 14.9 (7.79)
  Week 24: number analyzed (Participants) | 91
  Week 24 | 14.7 (8.10)

23. Secondary Outcome: Percentage Change From Baseline in Total IgG in the Overall Population
Description: Samples were collected predose, on the day of IMP administration.
Time Frame: Baseline and Weeks 1, 2, 3, 17, 19, 21, 23, and 24
Population: Pharmacodynamic (PD) Analysis Set: Safety analysis set including participants with at least one serum post dose PD measurement.
Measure: Mean (Standard Deviation); unit: percentage of total IgG
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 133 | 67
percentage of total IgG
  Week 1 | -33.64 (26.018) | 0.60 (14.065)
  Week 2: number analyzed (Participants) | 132 | 64
  Week 2 | -50.68 (34.973) | 10.31 (44.858)
  Week 3: number analyzed (Participants) | 131 | 64
  Week 3 | -56.80 (39.133) | 4.97 (28.484)
  Week 17: number analyzed (Participants) | 96 | 45
  Week 17 | -64.76 (11.478) | 1.27 (16.749)
  Week 19: number analyzed (Participants) | 98 | 51
  Week 19 | -60.98 (26.460) | 9.28 (44.989)
  Week 21: number analyzed (Participants) | 89 | 49
  Week 21 | -62.38 (15.176) | 4.62 (25.406)
  Week 23: number analyzed (Participants) | 92 | 49
  Week 23 | -62.45 (20.286) | 2.45 (21.271)
  Week 24: number analyzed (Participants) | 102 | 55
  Week 24 | -61.97 (18.200) | -0.36 (17.408)

24. Secondary Outcome: Number of Participants With Antiplatelet Antibodies in the Overall Population
Description: The antiplatelet antibody was positive if optical density value >0.129.
Time Frame: Weeks 7, 15, 23, and 24
Population: PD Analysis Set: Safety analysis set including participants with at least one serum post dose PD measurement and tested positive for antiplatelet antibodies at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 36 | 16
Participants
  Week 7: number analyzed (Participants) | 36 | 14
  Week 7 | 20 | 10
  Week 15: number analyzed (Participants) | 33 | 16
  Week 15 | 18 | 10
  Week 23: number analyzed (Participants) | 28 | 14
  Week 23 | 17 | 9
  Week 24: number analyzed (Participants) | 32 | 13
  Week 24 | 19 | 8

ADVERSE EVENTS:
Time Frame: Up to 35 weeks
Description: The total number of participants affected by other (not including serious) adverse events (AEs) include participants who experienced other AEs under the frequency threshold of 5%.
  SAF: All participants who received at least 1 dose or part of a dose.
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
All-Cause Mortality (participants affected / at risk) | 1/137 | 0/70
Serious Adverse Events (participants affected / at risk) | 14/137 | 10/70
Other Adverse Events (participants affected / at risk) | 130/137 | 65/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=137) | Placebo PH20 SC (N=70)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=137) | Placebo PH20 SC (N=70)
Anaemia (Blood and lymphatic system disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Gingival bleeding (Gastrointestinal disorders) | 14 | 10
Mouth haemorrhage (Gastrointestinal disorders) | 19 | 6
Oral blood blister (Gastrointestinal disorders) | 10 | 1
Fatigue (General disorders) | 8 | 0
Injection site bruising (General disorders) | 13 | 2
Injection site erythema (General disorders) | 9 | 2
Injection site haemorrhage (General disorders) | 14 | 14
Injection site pain (General disorders) | 8 | 2
Injection site rash (General disorders) | 7 | 1
Injection site reaction (General disorders) | 10 | 1
Vessel puncture site haemorrhage (General disorders) | 3 | 5
COVID-19 (Infections and infestations) | 18 | 6
Upper respiratory tract infection (Infections and infestations) | 12 | 6
Urinary tract infection (Infections and infestations) | 8 | 6
Contusion (Injury, poisoning and procedural complications) | 22 | 12
Blood urine present (Investigations) | 43 | 20
C-reactive protein increased (Investigations) | 3 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 8 | 3
Headache (Nervous system disorders) | 16 | 7
Haematuria (Renal and urinary disorders) | 32 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 15
Ecchymosis (Skin and subcutaneous tissue disorders) | 34 | 20
Petechiae (Skin and subcutaneous tissue disorders) | 34 | 19
Purpura (Skin and subcutaneous tissue disorders) | 15 | 11
Haematoma (Vascular disorders) | 7 | 3
Hypertension (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04687072/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04687072/SAP_001.pdf